CLINICAL TRIAL: NCT07357389
Title: VR for ICU Delirium Prevention
Brief Title: Virtual Reality for ICU Delirium Prevention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Devon Callahan, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004538
Record Dates: First submitted 2025-12-10; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: ICU Delirium
Keywords: ICU Delirium; Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard ICU delirium prevention (No Intervention)
- Study ICU Delirium Prevention and VR treatment (Experimental)
  Interventions: Device: Virtual Reality therapeutics

INTERVENTIONS:
Device: Virtual Reality therapeutics — Patients will receive daily VR sessions for up to 5 days in addition to regular delirium prevention measures in the ICU
  Arms: Study ICU Delirium Prevention and VR treatment

SUMMARY:
The purpose of this study is to evaluate whether daily exposure to immersive virtual reality (VR) can reduce the incidence of delirium in high-risk, non-intubated ICU patients. Participants will be randomized to either standard ICU care or standard care plus once-daily 15-minute VR sessions consisting of calming natural scenes, guided meditation, and music. The study population includes adult surgical ICU patients at Cedars-Sinai who are CAM-ICU negative at enrollment and possess at least one established risk factor for delirium. Outcomes will include the incidence and duration of delirium, ICU and hospital length of stay, feasibility of the VR intervention, and the frequency of adverse events. By targeting a high-risk population with an innovative non-pharmacologic therapy, this trial aims to generate data to support integration of VR into ICU delirium prevention protocols.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are currently admitted to the SICU at Cedars-Sinai Medical Center
* Expected ICU stay >48 hours
* Richmond Agitation Sedation Scale (RASS) score between -1 to +2.
* CAM-ICU negative
* 1≤ risk factor for delirium (Age ≥ 65 years old, history of cognitive impairment, sepsis, Sequential Organ Failure Assessment (SOFA) score >5, history of alcohol or benzodiazepine abuse, recent major surgery)

Exclusion Criteria:

* Unwilling and/or unable to participate
* Intubation of tracheostomy
* Self-reported history of severe motion sickness
* Inability to follow commands (e.g. severe aphasia, deafness, GCS<13)
* The presence of a facial/head deformity that will prohibit the wearing of a VR head mounted device (HMD
* Those that require corrective lenses -2.5 or stronger that cannot be corrected with contact lenses
* Having had a seizure in the past year
* Unable to understand the instructions or to consent to participation in the study.
* Those who are pregnant
* Hemodynamic instability (MAP<65 despite support)
* End-of-life care
* Severe agitation or delirium (i.e. CAM-ICU + screen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 822 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of ICU Delirium | From enrollment in the study until ICU discharge. Assessed Day 1 in the morning and evening for the duration of the ICU admission, up to 24 months from enrollment.
  Using the CAM-ICU assessment, patients will be evaluated for the development of ICU delirium

SECONDARY OUTCOMES:
Duration of ICU delirium | From the time of study enrollment until the time of discharge from the ICU, up to 24 months from enrollment.
  Number of days the patient experienced ICU delirium while admitted to the ICU
ICU-LOS | From time admitted to the ICU until discharge from the ICU, up to 24 months from enrollment.
  ICU length of stay
H-LOS | From time admitted to the hospital until discharge from the hospital, up to 24 months from enrollment.
  Hospital Length of stay
Acceptability by patients | From time enrolled in the study until the patient has completed the study interventions (either on discharge from the ICU or after 5 days of interventions, whichever comes first), from Day 1 until Day 5 after enrollment.
  Able to complete VR sessions as detailed in the study
Number of adverse events | Adverse events related to VR, such as nausea, dizziness, seizures, will be assessed from the time of enrollment in the study up until the time of discharge from the hospital, from time of enrollment on Day 1 until Day 5 after enrollment, if applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Devon S Callahan, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No